CLINICAL TRIAL: NCT05642403
Title: A Phase Ia Dose Escalation, Randomized, Double-Blinded, and Placebo- Controlled Clinical Study of Single Dose and Multiple Doses of XW001 Inhalation Solution in Healthy Adult Subjects
Brief Title: A Study of XW001 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SCW1201-3011
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-11

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — XW001

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SAD Cohort A XW001 (Active Comparator): Single inhalation of XW001
  Interventions: Drug: XW001
- SAD Cohort A placebo (Placebo Comparator): Single inhalation of placebo
  Interventions: Drug: Placebo
- MAD Cohort B XW001 (Active Comparator): Multiple inhalations of XW001
  Interventions: Drug: XW001
- MAD Cohort B placebo (Placebo Comparator): Multiple inhalations of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XW001 — Inhaled XW001
  Other Names: XW001 Inhalational solution
  Arms: MAD Cohort B XW001; SAD Cohort A XW001
Drug: Placebo — Matched inhaled placebo
  Other Names: Matched placebo Inhalational solution
  Arms: MAD Cohort B placebo; SAD Cohort A placebo

SUMMARY:
This is the first-in-human, single-center, randomized, double-blinded, placebocontrolled, single-dose and multiple-dose escalation Phase Ia study

DETAILED DESCRIPTION:
Single ascending dose (SAD), healthy participants will be randomized to receive a single inhalational dose of either XW001 or placebo in each of the planned SAD cohorts. Multiple ascending dose (MAD), healthy participants will be randomized to receive inhalational doses of XW001 or placebo in each of the planned MAD cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18-45 years (including both ends), male or female;
2. Body mass index (BMI) of 19.0-28.0 kg/m2 (including both ends);
3. Subjects who fully understand the trial objectives, have a basic understanding of the pharmacological effects and possible risks of the investigational drug, and voluntarily sign an informed consent form;
4. Subjects who can communicate well with the investigators, and understand and abide by the requirements of this study.

Exclusion Criteria:

1. (Screening period) Subjects participated in any drug clinical trial or used the investigational drug within 3 months prior to the trial;
2. (Screening period/admission) Subjects with a medical history of diseases in cardiovascular system, digestive system, endocrine system, urinary system, nervous system, hematological, immunological (including personal or family history of hereditary immunodeficiency), or metabolic abnormalities, etc., that are still considered as clinically significantly by the investigators.
3. (Screening period) Subjects with previously diagnosed chronic obstructive pulmonary disease (COPD), asthma, or other clinically significant lung diseases, or with a medical history of acute upper and lower respiratory infection requiring intravenous injection of antimicrobial drugs or other hospitalization treatment within the past 3 months;
4. (Screening period/admission) Subjects who had underwent a surgery that is considered affecting the pharmacokinetics(PK) behaviors of the drug by the investigator within 6 months prior to the trial;
5. Patients with positive endogenous interleukin 29 (IL-29) level (i.e., the test result in the screening period is higher than the lower limit of quantification);
6. Subjects with lung function abnormality (measured forced expiratory volume in one second #FEV1)/predicted FEV1 ≤ 80% or measured forced vital capacity (FVC)/predicted FVC ≤ 80%);
7. Subjects who are unable to complete the study for other reasons or are not suitable to participate in the trial as judged by the investigators.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Safety/tolerance endpoints | 28 Days for Cohort A and 42 Days for Cohort B
  Number and percentage of treatment emergent adverse events (TEAE) and serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Li, Principal Investigator — The Third Hospital of Changsha
Locations (1):
- The Third Hospital of Changsha, Changsha, Hunan, China